CLINICAL TRIAL: NCT06148350
Title: Regaining Balance and Quality of Life: The Impact of Frenkel's Exercises in Patients With Sub-Acute Ischemic Stroke-A Randomized Controlled Trial
Brief Title: Frenkel's Exercises for Sub-Acute Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al- Shifa Physiotherapy Institute /Clinic (Other)
Responsible Party: Principal Investigator, Muhammad Faisal, Mr. Muhammad Faisal, Al- Shifa Physiotherapy Institute /Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlShifa
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; Disability; Exercise; Balance; Quality of Life.
MeSH Terms: conditions — Ischemic Stroke; Stroke; Motor Activity | interventions — Stroke Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Frenkel's Exercise (Experimental): Frenkel's exercises spanned four weeks with distinct positions:
  Week 1: Recumbent position, focusing on heel sliding, knee, and hip movements. Week 2: Seated exercises, emphasizing leg elevation and standing from a chair. Week 3: Erect posture activities, including forward, sideways, and backward walking with diverse steps and turns.
  Week 4: Comprehensive exercises across all positions, emphasizing varied movements.
  Each exercise set included 8-10 repetitions with 1-2 minutes of rest.
  Interventions: Other: Stroke Rehabilitation
- Group B: Conventional Balance Exercises (Active Comparator): Structured program with 8-10 reps and 1-2 min rest:
  I. Strengthening: Targets hips, knees, and ankles-squats, lunges, leg presses. II. Weight-Shifting: Enhances balance with side-to-side, forward-backward steps.
  III. Trunk Stabilization: Improves core control-planks, crunches, twists. IV. Proprioception: Balance board exercises challenge spatial awareness, performed under physiotherapist supervision.
  Interventions: Other: Stroke Rehabilitation

INTERVENTIONS:
Other: Stroke Rehabilitation — Both the groups received interventions three days/week for 30-60 minutes for four weeks

SUMMARY:
This single-blinded, randomized controlled was aimed to compare the efficacy of Frenkel's and Conventional Balance Exercises in improving balance and quality of life in patients with subacute ischemic stroke. The participants of Group A received 'Frenkel's Exercises'. In contrast, Group B participants received 'Conventional Balance Exercise' interventions three days/week for 30-60 minutes for four weeks. The data was collected pre and post-treatment on the Berg Balance Scale and Stroke Specific-Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 35 to 75 years.
2. First-ever ischemic stroke and hemiparesis within 7 to 30 days of onset.
3. Reduced proprioception of the lower limb with a score of ≤12 on the NSA (kinesthetic and tactile sensation test),
4. Able to comprehend tasks and follow directions with a score of ≥21 points on the Mini-Mental State Examination (MMSE).
5. Able to independently perform standing motions for ≥1 minute.

Exclusion Criteria:

1. Patients with lower limb fractures within 6 months.
2. Severe pain.
3. Limited range of motion.
4. Cerebellar ataxia.
5. Medically unstable.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline
  The scale assesses dynamic balance skills with 14 items on a 5-point scale (0-4) and a total score of 56. It has a very high-reliability rating, with an ICC of 0.98. Participants who receive scores of 0 to 20 use wheelchairs, those who receive scores of 21 to 40 need aid or assistance, and those who receive scores of 41 or higher have independent gait.
Berg Balance Scale | After 4-weeks
  It has 14 items on a 5-point scale (0-4) and a total score of 56. It has a very high reliability rating, with an ICC of 0.98. Participants who receive scores of 0 to 20 use wheelchairs, those who receive scores of 21 to 40 need aid or assistance, and those who receive scores of 41 or higher have independent gait.
Stroke-Specific Quality of Life Scale | Baseline
  The scale measures the quality of life of participants. There are 49 items on the 5-point scale, with the lowest score being 49 and the highest being 245. The higher the quality of life, the lower the score. A Cronbach's alpha of 0.80 was reported as the test's reliability.
Stroke-Specific Quality of Life Scale | After 4-weeks
  The scale measures the quality of life of participants. There are 49 items on the 5-point scale, with the lowest score being 49 and the highest being 245. The higher the quality of life, the lower the score. A Cronbach's alpha of 0.80 was reported as the test's reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Shifa Physiotherapy Clinic Qasimabad Hyderabad, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No